CLINICAL TRIAL: NCT03477604
Title: A Clinical Evaluation of the MicroSTent® PeripherAl Vascular SteNt in Subjects With Arterial Disease Below the Knee (STAND)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Micro Medical Solution, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMS-001; NCT04025008 (obsolete NCT alias)
Record Dates: First submitted 2018-03-08; First posted 2018-03-26 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Below the knee; Stent
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MicroStent and Standard PTA (Experimental): Implant of the MicroStent peripheral vascular stent system for treatment of arterial lesions below the knee.
  Interventions: Device: MicroStent and Standard PTA
- Standard PTA (Active Comparator)
  Interventions: Device: Standard PTA

INTERVENTIONS:
Device: MicroStent and Standard PTA — Self-expanding stent and standard PTA balloon
  Arms: MicroStent and Standard PTA
Device: Standard PTA — Standard PTA balloon
  Arms: Standard PTA

SUMMARY:
Randomized multicenter clinical trial consisting of two arms; one arm treated with PTA plus the MicroStent® System and one arm treated with PTA alone. Purpose to evaluate the safety and effectiveness of using the MicroStent® Peripheral Vascular Stent System, hereafter referred to as the MicroStent® System, for the treatment of infrapopliteal lesions in subjects with peripheral arterial disease.

ELIGIBILITY:
General Inclusion Criteria:

1. Subject is a male or a non-pregnant female adult between the age of 21 and 90 years old.
2. Subject has documented clinical evidence of critical limb ischemia (CLI) in the target limb prior to the index procedure, with a Rutherford Classification score of 4-5.
3. The subject, or subject's designated legal representative, has been informed of the nature of the study and is willing to provide written informed consent.
4. Subject is willing to comply with all required follow-up visits.
5. Subject life expectancy is ≥1 year per the Principal Investigator.

   Angiographic Inclusion Criteria
6. Target vessel reconstitutes at or above the ankle with inline flow to at least one patent (<50% stenosis) inframalleolar outflow vessel.
7. Subject has a lesion, with ≥ 70% stenosis and ≤ 12.0 cm in length located at or distal to the tibial-peroneal trunk and above the tibiotalar joint; including the anterior tibial, posterior tibial or peroneal arteries.
8. Target lesion has a reference vessel diameter of 2.5 - 4.5 mm
9. The target lesion is able to be crossed with a guidewire to facilitate treatment with the randomized device.

General Exclusion Criteria:

1. Subject had a prior or has a planned index limb amputation above the ankle.
2. Subject has a wound/ulcer on the forefoot with a surface area >4cm² or osteomyelitis involving the calcaneus bone.
3. Subject is pregnant, plans to become pregnant, or is nursing.
4. Subject has clinical conditions that severely inhibit X-ray or duplex ultrasound visualization (e.g. body habitus).
5. Subject has a history of hypercoagulation/clotting disorders or acute thrombosis.
6. Subject has allergy to iodinated contrast media that cannot be adequately managed with medication.
7. Subject is in acute renal failure.
8. Subject has an active systemic infection.
9. Subject is participating in another research study involving an investigational device, biologic, or drug that has not completed the primary endpoint at the time of randomization/enrollment.
10. Subject has other comorbidities that - in the opinion of the investigator - preclude them from receiving study treatment and/or from completing the required study follow-up assessments.
11. Subject presents with acute limb ischemia or acute thrombosis of the target limb.
12. Subject has experienced myocardial infarction, thrombolysis, or angina less than 30 days prior to the index procedure.
13. Subject had a stroke within 3 months of index procedure.

    Angiographic exclusion criteria
14. Failure to successfully treat clinically significant inflow lesions in the ipsilateral iliac, femoral, or popliteal arteries. Successful treatment is defined as obtaining ≤30% residual stenosis with no major procedural complications (e.g embolism).
15. Failure to successfully treat significant non-target infra-popliteal lesions. Successful treatment is defined as obtaining ≤30% residual stenosis with no major procedural complications (e.g. embolism).
16. Target lesion is within a previously placed stent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Patency of the target lesion | up to 6 months after randomization
  Primary patency defined as freedom from target lesion occlusion with no clinically driven target lesion reintervention, or major amputation.
Freedom from perioperative death | up to 30 days after randomization
  Freedom from perioperative death
Freedom from major adverse limb event | up to 6 months after randomization
  Freedom from major adverse limb event

SECONDARY OUTCOMES:
Freedom from major amputation above the ankle | up to 6 months after randomization
  Freedom from major amputation (above the ankle)
Reduction in size of ischemic leg/foot ulcers | up to 6 months after randomization
  Reduction in size of ischemic leg/foot ulcers
Freedom from major adverse limb event | From date of randomization until the date of death from any cause assessed up to 36 months
  Freedom from major adverse limb event
Frequency and severity of serious adverse events and device and procedure related adverse events | From date of randomization until the date of death from any cause assessed up to 36 months
  Frequency and severity of serious adverse events and device and procedure-related adverse events at any time during the study.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Cardiovascular Associates of the Southeast, Birmingham, Alabama
  - Copper State Vascular, Mesa, Arizona
  - St. Helena Hospital, St. Helena, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Palm Vascular, Fort Lauderdale, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - FHV Health, Leesburg, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Advent Health Sebring, Sebring, Florida
  - Vascular Institute of the Midwest, Davenport, Iowa
  - Cardiovascular Institute of the South, Houma, Louisiana
  - University of Maryland - Baltimore, Baltimore, Maryland
  - Advanced Cardiac and Vascular Amputation Prevention Centers, Grand Rapids, Michigan
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - North Jersey Vascular Center, Clifton, New Jersey
  - AMI Vascular Institute, Galloway, New Jersey
  - US Cardiovascular, Jefferson Hills, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Cardiology Consultants, Spartanburg, South Carolina
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - AZH/WAVE Vascular Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No